CLINICAL TRIAL: NCT03130244
Title: A Trial for a Procedure for Duodenum to Ileal Diversion to Treat Type 2 Diabetes
Brief Title: Procedure for Duodenum to Ileal Diversion to Treat Type 2 Diabetes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GI Windows, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GIW 16-001
Record Dates: First submitted 2017-04-21; First posted 2017-04-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Type 2 Diabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Device Placement (Active Comparator): The patients in this arm will receive the Magnet Anastomosis System and an anastomosis will be created.
  Interventions: Device: Magnet Anastomosis System; Drug: Best Medical Management
- Control (No Intervention): The patients in this arm will receive the best medical management.

INTERVENTIONS:
Device: Magnet Anastomosis System — The MAS will be placed using an endoscope in the duodenum and and laparoscopically into ileum. A compression anastomosis will be created in each of the patients and the diversion of enteral flow from the duodenum to ileum treats Type 2 diabetes.
  Other Names: MAS
  Arms: Device Placement
Drug: Best Medical Management — The best medical management for the patients in this arm will be decided by the endocrinologist based on protocol parameters.
  Other Names: No other intervention
  Arms: Device Placement

SUMMARY:
Study will monitor changes in HbA1c for subjects in Intervention arm vs control arm.

DETAILED DESCRIPTION:
Randomized, Single-Center, Parallel-group, Open-label Pilot Study to Evaluate the Safety and Effectiveness of the GI Windows Magnet Anastomosis System (MAS) When Used to Create a Dual-path Enteral Diversion Compared with Medical Therapy Alone To Effect Glycemic Control in Obese Patients with Type 2 Diabetes Mellitus (T2DM)

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) 30 to 50.
* Subject Type 2 Diabetes Criteria:

  1. T2DM diagnosis ≥6 months but < 10 years
  2. On 1 or more oral diabetes medications (with one at the minimum recommended therapeutic dose)
  3. Hemoglobin A1C (HbA1c) between and including 6.5 and 10.0% (58 mmol/mol to 86 mmol/mol) at time of enrollment and has had a stable HbA1c over a 3-month period (i.e., <0.3% reduction)
  4. Stable medication regimen (i.e., no change in diabetes medications) for at least 3 months prior to Screening Visit.
* If subject has obesity-related comorbidities such as hypertension, dyslipidemia, and sleep apnea, these comorbidities must be well-controlled.
* Able to understand and sign informed consent document
* Has primary care physician and/or endocrinologist who follows patient for all comorbid conditions

Exclusion Criteria:

* Known or suspected allergy to nickel or titanium or Nitinol
* Type 1 Diabetes
* Use of injectable insulin
* Uncontrolled T2DM Fasting glucose ≥ 200 mg/dl (11.1 mmol/L)
* Probable insulin production failure, defined as fasting serum C Peptide <1 ng/mL (0.3 nmol/l)
* Any documented conditions for which endoscopy/colonoscopy would be contraindicated.
* Contraindication to general anesthesia
* Congenital or acquired anomalies of the GI tract, including atresias, stenosis or malrotation.
* Any previous major surgery on the stomach (excluding sleeve gastrectomy), duodenum, hepatobiliary tree (excluding gallbladder), pancreas or right colon.
* Previous technically difficult or failed colonoscopy or endoscopy
* If on metformin, history of polycystic ovarian syndrome (PCOS)
* Unable or unwilling to perform home blood glucose monitoring
* History of or suspected gastrointestinal disease (e.g. cirrhosis, inflammatory bowel disease)
* Diagnosis of active malignancy (i.e. not in remission) with the exception of squamous or basal cell carcinoma of the skin
* Previous surgical or endoscopic treatment for obesity including but not restricted to intragastric balloons, endoscopic suturing or stapling procedures, malabsorptive sleeves.
* Specific genetic or hormonal cause of obesity (e.g. Prader-Willi syndrome)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Mean change in HbA1c | 12 months
  The primary effectiveness endpoint is Mean change in HbA1c from baseline

SECONDARY OUTCOMES:
Mean change in Weight | 12 months
  12 month weight loss measured as a percent of total body weight loss and excess weight loss (using the BMI method) as well as weight/BMI change from baseline
Proportion of subjects achieving remission | 12 months
  Proportion of subjects experiencing diabetes remission and/or partial remission at 12 months (as defined by the American Diabetes Association)
Mean change in diabetes medication | 12 months
  Change in diabetes medication requirements from baseline to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf H Buxhoeveden, Principal Investigator — Bariatric Surgeon at Hospital Aleman
Locations (1):
- Aleman Hospital, Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No